CLINICAL TRIAL: NCT04142203
Title: 23 Hour Surgical Model in a Tertiary Hospital: Evaluation From Patient and Organisational Perspective
Brief Title: Implementation of 23 Hour Surgery Model in a Tertiary Hospital
Acronym: Herko
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KUH507A030
Record Dates: First submitted 2019-10-17; First posted 2019-10-29 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-02

CONDITIONS: Ambulatory Surgery; Laparoscopy; Shoulder Impingement Syndrome; Ovarian Cysts; Cholecystolithiasis; Appendicitis; Gynecologic Surgical Procedures; Ambulatory Surgical Procedures; Neurosurgery
Keywords: 23 h surgery; postoperative recovery; outcome; patient satisfaction; postoperative pain; analgesic; oxycodone; multimodal pain management; extended day surgery
MeSH Terms: conditions — Shoulder Impingement Syndrome; Ovarian Cysts; Cholecystolithiasis; Appendicitis; Patient Satisfaction; Pain, Postoperative | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 23 h surgery: Adult patients who were treated in 23 h surgical unit
  Interventions: Other: 23 h surgery

INTERVENTIONS:
Other: 23 h surgery — Patients were treated in 23 surgical unit

SUMMARY:
Extended day surgery or 23 h surgery (23-hour surgery) is a surgical model where patients arrive to the hospital from home at the day of surgery, are operated and recover in a 23 h surgery unit. 23H surgery units are usually situated near postoperative recovery unit. THe 23 H surgical model was implemented in Kuopio University Hospital 2015 and between May 2017-May 2018 patients were recruited in the present prospective follow up cohort study. Patients were informed and they gave their informed consent. The patients were contacted two weeks after the study and details of their recovery were asked.

DETAILED DESCRIPTION:
Extended day surgery or 23 h surgery is a surgical model where patients arrive to the hospital from home at the day of surgery, are operated and recover in a 23 h surgery unit. 23H surgery units are usually situated near postoperative recovery unit. THe 23 H surgical model was implemented in Kuopio University Hospital 2015 and between May 2017-May 2018 patients were recruited in the present prospective follow up cohort study. Patients were informed and they gave their informed consent. The patients were contacted two weeks after the study and details of their recovery were asked. Satisfaction to the care in 23 h unit and surgical process, were asked. Amount of readmissions, reoperations, contacts to health care professionals and adverse events are recorded.

Detailed information about intensity of pain, analgesic need and use in the hospital was recorded and pain interference in daily life for short term recovery period was asked.

ELIGIBILITY:
Inclusion Criteria:

* adult
* gave informed consent

Exclusion Criteria:

* no informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing 23 h surgery
Sampling Method: Non-Probability Sample
Enrollment: 993 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Amount of patients discharged from the hospital until 10 am at the first postoperative day | Postoperative day 1
  The amount of patients discharged from hospital by the first postoperative day 10 am
Pain intensity postoperatively | Postoperative day 1
  Pain intensity after surgery for the first 24 hours
Analgesic consumption postoperatively | Postoperative day 1
  Amount of different analgesics consumed during the 24 h period postoperatively

SECONDARY OUTCOMES:
30 days readmission rate | one month after surgery
  How many patients are admitted to hospital within 30 postoperative days
30 days reoperation rate | one month after surgery
  How many patients are reoperated within 30 postoperative days
Number of adverse events during 14 postoperative days | 14 days after surgery
  Amount of adverse events after surgery within 14 postoperative days
Contact to health care during 14 postoperative days | 14 days afte surgery
  Number of contacts to health care within 14 postoperative days
Patient satisfaction to care in 23 hours process | 14 days after surgery
  Scale 0-7 (0= not satisfied, 7 =very satisfied), the higher score the better result
Proportion of patients having pain postoperatively | Two weeks postoperatively
  Amount of patients who had pain still two weeks after surgery
Postoperative pain interference after 23 h surgery | two weeks postoperatively
  Patient assessed pain interference in daily activities up to 2 weeks after surgery
Analgesic use after 23 h surgery | Two weeks postoperatively
  amount of patients using analgesics two weeks after surgery

OTHER OUTCOMES:
Adverse events after 23 h surgery | two weeks after surgery
  Adverse events after 23 h surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ulla-Maija Ruohoaho, MD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Isokaanta S, Ruohoaho UM, Anttila M, Kokki H, Sintonen H, Toroi P, Kokki M. Resilience, pain, and health-related quality of life in gynecological patients undergoing surgery for benign and malignant conditions: a 12-month follow-up study. BMC Womens Health. 2022 Aug 16;22(1):345. doi: 10.1186/s12905-022-01923-7. PMID 35974326
- [Derived] Ruohoaho UM, Aaltomaa S, Kokki H, Anttila M, Kokki M. Patient functional recovery after a 23-h surgery - a prospective, follow-up study. Langenbecks Arch Surg. 2022 Aug;407(5):2133-2142. doi: 10.1007/s00423-022-02502-y. Epub 2022 Apr 6. PMID 35384504
- [Derived] Ruohoaho UM, Toroi P, Hirvonen J, Aaltomaa S, Kokki H, Kokki M. Implementation of a 23-h surgery model in a tertiary care hospital: a safe and feasible model with high patient satisfaction. BJS Open. 2020 Jun;4(3):391-399. doi: 10.1002/bjs5.50267. Epub 2020 Feb 28. PMID 32109004